CLINICAL TRIAL: NCT01670968
Title: The Effect of Antiretroviral Therapy and HIV on Reverse Cholesterol Transport in Blood( HIV Reverse Cholesterol Transport Study- HIV RCTS)
Brief Title: HIV Reverse Cholesterol Transport Study
Acronym: HIV RCTS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College Dublin (Other)
Collaborators: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Patrick Mallon, Associate Dean for Research and Innovation UCD School of Medicine and Medical Sciences, Consultant Infectious Diseases Physician, University College Dublin
Other Study IDs: HIV RCTS
Record Dates: First submitted 2012-08-18; First posted 2012-08-23 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: HIV; Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary Objective:

To examine changes in expression of genes [particularly ABCA1 and SREBP2] involved in reverse cholesterol transport (RCT) in monocytes from HIV-infected subjects starting antiretroviral therapy and the different effect of NNRTI and PI based regimens

Secondary Objective:

To examine changes in monocyte intracellular cholesterol content in HIV-infected subjects starting antiretroviral therapy and the different effect of NNRTI and PI based regimens

DETAILED DESCRIPTION:
HIV infection is associated with low HDL-cholesterol, an independent risk-factor for cardiovascular disease (CVD). NNRTI-based HAART increases HDL-c, with nevirapine shown to increase production of its major apolipoprotein ApoA-I. In contrast, initiation of PI-based HAART leads to persistently low HDL-c despite a reduction in HIV RNA and immunologic recovery.

HDL-c is formed through reverse cholesterol transport (RCT), the process where cholesterol is transferred from intracellular pools to circulating lipoproteins which are then eliminated by the liver. Accumulation of intracellular cholesterol in cells such as macrophages and their precursor (circulating monocytes) has been implicated in atherogenesis.

In vitro data suggests the HIV protein Nef directly interferes with cellular proteins involved in RCT such as ATP-binding cassette transporter A1 (ABCA1) in monocyte-derived macrophages. ABCA1 expression is controlled by peroxisome proliferator-activated receptor gamma (PPARG) and the intracellular cholesterol sensor sterol regulatory element binding protein 2 (SREBP2). In adipose tissue it is known that PI treatment downregulates SREBP and PPARG expression.

Preliminary work in the investigators lab has reproduced these findings in monocytes in untreated HIV infection in vivo and demonstrated relationships between gene expression for ABCA1, SREBP2, monocyte intracellular cholesterol and circulating lipoproteins. These early data suggest that defects in RCT determine intracellular cholesterol levels in HIV-infected subjects whereas increased LDL-c is a greater determinant of intracellular cholesterol in HIV negative subjects. This suggests a potentially pivotal role for RCT abnormalities in low HDL-c, increased intracellular cholesterol and atherogenesis in HIV infection.

The investigator's aim to examine the impact of initiation of ART with either PI or NNRTI on RCT in circulating monocytes in vivo and how this impact correlates with changes in amount and size of circulating HDL-c.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* HIV-infected
* Not currently on antiretroviral therapy (>6/12), but about to start

Exclusion Criteria:

* On lipid lowering medication (statin / fibrate / niacin)
* HCV Ab+

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals starting antiretroviral therapy at the Mater Misericordiae University Hospital, Dublin, and Chelsea and Westminister Hospital, London
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2020-05 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Change in ABCA1 mRNA expression in monocytes | June 2013

CONTACTS AND LOCATIONS:
Overall Officials: Patrick WG Mallon, FRACP FRCPI PhD, Principal Investigator — HIV Molecular Research Group, UCD School of Medicine and Medical Sciences. Department of Infectious Diseases, Mater Misericordiae University Hospital and Mater Private Hospital
Locations (1):
- Chelsea & Westminster Hospital, London, United Kingdom